CLINICAL TRIAL: NCT02546232
Title: Improved Breast Cancer Therapy (I-BCT-1) in the Neoadjuvant and Metastatic Setting: A Phase 2 Clinical Trial Protocol Studying Biological Rationale for the Optimal Selection of Treatment Regimens
Brief Title: Improved Breast Cancer Therapy (I-BCT-1) in the Neoadjuvant and Metastatic Setting
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Olav Engebraaten, Consultant oncologist / Associate professor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I-BCT-1
Record Dates: First submitted 2015-08-11; First posted 2015-09-10 (Estimated); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
Keywords: locally advanced breast cancer; metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Paclitaxel 80 mg/m2 weekly for 12 weeks, thereafter current standard chemotherapy for 12 weeks
  Interventions: Drug: Paclitaxel
- Additional therapy (Experimental): Carboplatin AUC 6 (area under curve; mg/ml/min) once every 3 weeks, for 12 weeks.
  Paclitaxel 80 mg/m2 weekly for 12 weeks, thereafter current standard chemotherapy for 12 weeks
  Interventions: Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Carboplatin — Chemotherapy
  Arms: Additional therapy
Drug: Paclitaxel — Chemotherapy
  Other Names: Taxol

SUMMARY:
The purpose of the study is to investigate the molecular biology of the tumor in relation to treatment response to chemotherapy, in particular paclitaxel compared to the combination paclitaxel and carboplatin. The study is carried out in two different, separate cohorts:

Cohort I: Patients with large primary breast cancer (> 2.0 cm) including locally advanced disease, are treated with weekly paclitaxel for 12 weeks, before continuing on anthracycline containing regimen for another 12 weeks before surgery. Patient are randomized 1:1 to receive carboplatin in addition to paclitaxel for the first 12 weeks of the treatment.

Cohort II: Patients with metastatic disease, available for biopsies before and during therapy are included to receive paclitaxel for 24 weeks. Patients are randomized 1:1 to receive paclitaxel alone or paclitaxel in combination with carboplatin.

DETAILED DESCRIPTION:
High-throughput methods in molecular biology have revealed considerable alterations in the breast cancer genome, transcriptome and proteome with extensive heterogeneity between tumors, potentially explaining the large variation in response to treatment. Classification of breast cancer can be based on such molecular alterations, and have shown to be of clinical relevance. Studies on how genome-wide mRNA (messenger ribonucleic acid) /miRNA (microRNA) expression, copy number alterations (CNAs) and DNA methylation, in addition to the detection of circulating tumor DNA could be used to improve prognostication and aid in therapy decision are highly needed. This project includes a phase II clinical trial where patients will be randomized to treatment with standard anthracycline- and taxane containing chemotherapy with or without the addition of carboplatin. The study aims to include patients in two cohorts as described, with large primary breast cancer (cohort I - 150 patients) and patients with metastatic disease (cohort II - 60 patients). Essential for the study is the mandatory tissue samples for comprehensive molecular analyses to identify markers of response.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained prior to any study-specific procedure
2. Female or male age ≥ 18 years
3. Able to comply with the protocol
4. Histologically or cytologically confirmed, HER2 (human epidermal growth factor 2) -negative, men or women with breast adenocarcinoma
5. WHO performance status ≤ 2
6. Adequate hematological function Absolute neutrophil count (ANC) ≥1.0 x 109/L AND Platelet count ≥100 x 109/L AND Hemoglobin ≥ 10 g/dL (may be transfused to maintain or exceed this level)
7. Adequate liver function Total bilirubin <1.5 x upper limit of normal (ULN) AND AST (aspartate aminotransferase), ALT (alanine aminotransferase) <2.5 x ULN (in cohort I); AST, ALT <5 x ULN (in cohort II)
8. Adequate renal function Serum creatinine ≤1.25 x ULN (and if measured: Creatinine clearance within normal reference values)
9. Women should not be pregnant or breast-feeding. Women with an intact uterus (unless amenorrhoeic for the last 24 months and premenopausal levels of FSH (follicle stimulating hormone), LH (luteinizing hormone) and oestradiol) must have a negative serum pregnancy test within 28 days prior to inclusion into the study.

Exclusion Criteria:

1. Previous chemotherapy treatment for localized breast cancer less than 24 months before inclusion into study (cohort I) or metastatic breast cancer treated with taxane (cohort II).
2. Other earlier or concomitant carcinoma less than five years prior to the breast cancer diagnosis, except for basal cell carcinoma, in situ cervix cancer or breast cancer
3. Clinically significant (i.e. active) cardiovascular disease for example cardiovascular accident (≤6 months before enrolment), myocardial infarction (≤6 months before enrolment), unstable angina, congestive heart failure (CHF) NYHA (New York Heart Association) Class ≥II, serious cardiac arrhythmia requiring medication during the study, which might interfere with regularity of the study treatment, or not controlled by medication
4. Treatment with any other investigational agent, or participation in another clinical intervention trial within 21 days prior to enrolment
5. Evidence of any other disease, neurological or metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or puts the patient at high risk for treatment-related complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment response: Cohort I - pCR (pathologic complete response), Cohort II - CR (complete response), PR (partial response), SD (stable disease), PD (progressive disease) | 24 weeks
  The primary objective of the study is to determine the molecular (DNA, RNA, protein and metabolic) changes in the tumors with reference to the obtained therapeutic response in the different treatment arms.

SECONDARY OUTCOMES:
Circulating tumor-DNA in plasma | 24 weeks
  Treatment induced changes and characteristics of circulating tumor DNA compared to tumor response
Fatigue (patient reported by standardized questionnaire) | 24 weeks
  Course of fatigue and predictors of chronic fatigue in the treatment arms.

CONTACTS AND LOCATIONS:
Overall Officials: Olav Engebraaten, MD, PhD, Principal Investigator — Department of Oncology, Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No